CLINICAL TRIAL: NCT01321372
Title: A Prospective, Observational Analysis of Voriconazole (VOR) Therapeutic Drug Concentration Monitoring, Pharmacogenomics and Clinical Outcome Correlations in High-risk Hematology Patients at Princess Margaret Hospital
Brief Title: An Observational Analysis of Voriconazole Therapeutic Drug Concentration Monitoring, Pharmacogenomics and Clinical Outcome Correlations in High-risk Hematology Patients
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: PMH-VOR
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hematology patients are at high risk for invasive fungal infection (IFI) and are being treated with voriconazole (VOR) at Princess Margaret Hospital (PMH). It is critical that patients' serum drug levels are within therapeutic ranges when undergoing treatment. The primary objective of this study is to determine whether clinical responses (complete/partial/failure) directly correlate with patients' blood VOR drug levels.

In patients whose disease progression is associated with inadequate voriconazole (VOR) drug levels, serum drug level determination can allow for dose adjustment, thereby preventing disease progression. Patients who are extensive metabolizers may have subtherapeutic VOR levels leading to treatment failure whereas, poor metabolizers may have high drug levels that cause toxicity. Isoenzyme such as CYP2C19 exhibits genetic polymorphism. Genotyping tests can also be helpful in determining patient risk subjecting to extreme spectrum of drug levels.

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia (including myelogenous and lymphocytic) patients for remission induction chemotherapy, reinduction chemotherapy and consolidation chemotherapy whose antifungal treatment include voriconazole.
* Patients have been subscribed voriconazole for probable or proven fungal infections by microbiological/cytohistological evidence from fine needle aspirate or bronchoalveolarlavage means.
* Patients will also have imaging positive from lose dose CT results depicting halo signs or crescent signs suggestive of invasive fungal infections.
* Patients must be able to tolerate oral intake of medications.

Exclusion Criteria:

* Patients unable to tolerate oral administration with any combinations of severe mucositis (> or = grade 3), nausea/vomiting (> or = grade 3), diarrhea (> or =grade 2), neutropenic enterocolitis (> or = grade3).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute leukemia (including myelogenous and lymphocytic) patients for remission induction chemotherapy, reinduction chemotherapy and consolidation chemotherapy whose antifungal treatment includes voriconazole.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-06; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine whether clinical responses (complete/partial/failure) directly correlate with patients' blood voriconazole levels. | 4 years
  The primary outcome measure is defined by the following endpoints:
  1. abefrile for at least 48 hours
  2. no breakthrough fungal infection
  3. resolution or improvement of radiological findings

SECONDARY OUTCOMES:
The secondary objective of this study will focus on clinical toxicity, organ involvement and survival. | 4 years
  The secondary outcome of the study is defined as resolution of renal or hepatic dysfunction and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Seki, P.Ph, PharmD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada